CLINICAL TRIAL: NCT01329978
Title: The ATOMIC Study: A Multicenter, Open-label, Randomized, Duration Finding Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics Following Oral Administration of PSI-7977 in Combination With Pegylated Interferon and Ribavirin in Treatment-Naive Patients With Chronic HCV Infection Genotype 1,4, 5, or 6
Brief Title: Sofosbuvir With Pegylated Interferon and Ribavirin Hepatitis C Virus (HCV) Genotypes 1,4,5,6
Acronym: ATOMIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P7977-0724
Record Dates: First submitted 2011-03-30; First posted 2011-04-06 (Estimated); Results first posted 2014-05-26 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-04

CONDITIONS: Hepatitis C, Chronic
Keywords: Hepatitis C; HCV; Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — Sofosbuvir; Ribavirin; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- SOF+PEG+RBV 12 weeks (Experimental): Participants were randomized to receive sofosbuvir+PEG+RBV for 12 weeks.
  Interventions: Drug: Sofosbuvir; Drug: RBV; Drug: PEG
- SOF+PEG+RBV 24 weeks (Experimental): Participants were randomized to receive sofosbuvir+PEG+RBV for 24 weeks.
  Interventions: Drug: Sofosbuvir; Drug: RBV; Drug: PEG
- SOF+PEG+RBV 12 week/Rerandomization Group (Experimental): Participants were randomized to receive sofosbuvir+PEG+RBV for 12 weeks, then were rerandomized to receive sofosbuvir only or sofosbuvir+RBV for 12 additional weeks.
  Interventions: Drug: Sofosbuvir; Drug: RBV; Drug: PEG

INTERVENTIONS:
Drug: Sofosbuvir — Sofosbuvir (SOF) administered as a 400 mg tablet orally once daily
  Other Names: Sovaldi®; GS-7977; PSI-7977
Drug: RBV — Ribavirin (RBV) tablets administered orally in a divided daily dose according to package insert weight-based dosing recommendations (< 75kg = 1000 mg and ≥ 75 kg = 1200 mg)
  Other Names: Copegus®
Drug: PEG — Pegylated interferon alfa-2a (PEG) 180 μg administered once weekly by subcutaneous injection
  Other Names: Pegasys®

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and efficacy of sofosbuvir (GS-7977; PSI-7977) administered in combination with pegylated interferon and ribavirin (PEG/RBV) in treatment-naive patients with HCV genotypes 1,4,5,6, or indeterminate genotype.

ELIGIBILITY:
Inclusion Criteria:

* Males and females with Chronic Hepatitis C (HCV) Genotype 1,4,5,6, or indeterminate
* Naive to previous HCV treatment

Exclusion Criteria:

* Positive for HBsAg, anti-HBc IgM Ab, or anti-HIV Ab
* History of any other clinically significant chronic liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2011-03; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert H. Hyland, DPhil, Study Director — Gilead Sciences
Locations (46):
- United States (44):
  - Alabama Liver and Digestive Specialist, Montgomery, Alabama
  - Clopton Clinic, Jonesboro, Arkansas
  - Advanced Clinical Research Institute, Anaheim, California
  - Providence Clinical Research, Burbank, California
  - Southern California Liver Centers, Coronado, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - eStudy Site, Oceanside, California
  - Desta Digestive Disease Medical Center, San Diego, California
  - Medical Associates Reseach Group, San Diego, California
  - Kaiser Permanente Hepatology Research, San Diego, California
  - University of Colorado Denver Transplant Center and Hepatology Clinic, Aurora, Colorado
  - South Denver Gastreoenterology, Englewood, Colorado
  - Pointe West Infectious Disease, Bradenton, Florida
  - Avail Clinical Research, DeLand, Florida
  - University of Florida College of Medicine, Gainesville, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Internal Medicine Specialists, Orlando, Florida
  - Advanced Research Institute, Trinity, Florida
  - South Florida Center of Gastroenterology, Wellington, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Gastrointestinal Specialists of Georgia, Marietta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Investigative Clinical Research, Annapolis, Maryland
  - Clinical Associates Research, Reisterstown, Maryland
  - Beth Israel Deconess Medical Center, Boston, Massachusetts
  - U Mass Memorial Medical Center, Worcester, Massachusetts
  - Henry Ford Health System, Novi, Michigan
  - St. Louis University Gastroenterology and Hepatology Clinical Research, St Louis, Missouri
  - University of New Mexico Health Science Center, Albuquerque, New Mexico
  - North Shore University Hospital, Manhasset, New York
  - Concorde Medical Group, New York, New York
  - New York Presbyterian Hospital, New York, New York
  - Mt. Sinai Medical Center, New York, New York
  - Asheville Gastroenterology Associates, Asheville, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Columbia Gastroenterology Associates, Columbia, South Carolina
  - North Texas Research Institute, Arlington, Texas
  - Central Texas Cinical Research, Austin, Texas
  - Baylor University, Dallas, Texas
  - Baylor/ St. Luke's Advanced Liver Therapy, Houston, Texas
  - Alamo Medical Research, San Antonio, Texas
  - Digestive and Liver Disease Specialist, Norfolk, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
- Puerto Rico (2):
  - University Of Puerto Rico, San Juan, Puerto Rico
  - Fundacion de Investigacion de Diego, San Juan, Puerto Rico

REFERENCES:
- [Derived] Lawitz E, Poordad FF, Pang PS, Hyland RH, Ding X, Mo H, Symonds WT, McHutchison JG, Membreno FE. Sofosbuvir and ledipasvir fixed-dose combination with and without ribavirin in treatment-naive and previously treated patients with genotype 1 hepatitis C virus infection (LONESTAR): an open-label, randomised, phase 2 trial. Lancet. 2014 Feb 8;383(9916):515-23. doi: 10.1016/S0140-6736(13)62121-2. Epub 2013 Nov 5. PMID 24209977
- [Derived] Kowdley KV, Lawitz E, Crespo I, Hassanein T, Davis MN, DeMicco M, Bernstein DE, Afdhal N, Vierling JM, Gordon SC, Anderson JK, Hyland RH, Dvory-Sobol H, An D, Hindes RG, Albanis E, Symonds WT, Berrey MM, Nelson DR, Jacobson IM. Sofosbuvir with pegylated interferon alfa-2a and ribavirin for treatment-naive patients with hepatitis C genotype-1 infection (ATOMIC): an open-label, randomised, multicentre phase 2 trial. Lancet. 2013 Jun 15;381(9883):2100-7. doi: 10.1016/S0140-6736(13)60247-0. Epub 2013 Mar 15. PMID 23499440

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in a total of 42 study sites in the United States. The first participant was screened on 23 March 2011. The last participant observation was on 27 August 2012.
Pre-assignment Details: 589 participants were screened and 332 were randomized and treated, and comprise the Safety Analysis Set.
Groups:
- SOF+PEG+RBV 12 Weeks: Participants were randomized to receive sofosbuvir (SOF) 400 mg+pegylated interferon alfa-2a (PEG) 180 µg+ribavirin (RBV) 1000-1200 mg for 12 weeks.
- SOF+PEG+RBV 24 Weeks: Participants were randomized to receive SOF 400 mg+PEG 180 µg+RBV 1000-1200 mg for 24 weeks.
- SOF+PEG+RBV 12 Week/Rerandomization Group: Participants were randomized to receive SOF 400 mg+PEG 180 µg+RBV 1000-1200 mg for 12 weeks, then were rerandomized to receive SOF monotherapy or SOF+RBV for 12 additional weeks.
- SOF Rerandomization Group: This group includes participants in the SOF+PEG+RBV 12 week/Rerandomization Group who were rerandomized to receive SOF 400 mg monotherapy for 12 additional weeks.
- SOF+RBV Rerandomization Group: This group includes participants in the SOF+PEG+RBV 12 week/Rerandomization Group who were rerandomized to receive SOF 400 mg+RBV 1000-1200 for 12 additional weeks.
Period: Sofosbuvir+PEG+RBV Treatment Period
Arm/Group | SOF+PEG+RBV 12 Weeks | SOF+PEG+RBV 24 Weeks | SOF+PEG+RBV 12 Week/Rerandomization Group | SOF Rerandomization Group | SOF+RBV Rerandomization Group
Started | 52 | 125 | 155 | 0 | 0
Completed | 48 (Participants in this group were not re-randomized for further treatment) | 112 (Participants in this group were not re-randomized for further treatment) | 150 (150 participants were re-randomized after 12 weeks of treatment.) | 0 | 0
Not Completed | 4 | 13 | 5 | 0 | 0
Not completed — Adverse Event | 1 | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 8 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 3 | 0 | 0
Not completed — Subject Was Incarcerated | 0 | 1 | 0 | 0 | 0
Not completed — Subject Moved Out of State | 0 | 1 | 0 | 0 | 0
Period: Rerandomization Treatment Period
Arm/Group | SOF+PEG+RBV 12 Weeks | SOF+PEG+RBV 24 Weeks | SOF+PEG+RBV 12 Week/Rerandomization Group | SOF Rerandomization Group | SOF+RBV Rerandomization Group
Started | 0 | 0 | 0 | 75 (This group includes participants rerandomized from the SOF+PEG+RBV 12 week/Rerandomization Group.) | 75 (This group includes participants rerandomized from the SOF+PEG+RBV 12 week/Rerandomization Group.)
Completed | 0 | 0 | 0 | 70 | 71
Not Completed | 0 | 0 | 0 | 5 | 4
Not completed — Lost to Follow-up | 0 | 0 | 0 | 5 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who were randomized and received at least 1 dose of study drug
Groups:
- SOF+PEG+RBV 12 Weeks: Participants were randomized to receive SOF 400 mg+PEG 180 µg+RBV 1000-1200 mg for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | SOF+PEG+RBV 12 Weeks | SOF+PEG+RBV 24 Weeks | SOF+PEG+RBV 12 Week/Rerandomization Group | Total
Number analyzed (Participants) | 52 | 125 | 155 | 332
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (9.8) | 50 (11.0) | 50 (10.8) | 50 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 52 | 49 | 118
  Male | 35 | 73 | 106 | 214
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 26 | 31 | 67
  Not Hispanic or Latino | 42 | 99 | 124 | 265
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 2 | 17 | 16 | 35
  Not Black | 50 | 108 | 139 | 297
Hepatitis C Virus (HCV) genotype [Number; unit: participants] — There are variations of HCV which are all similar enough to be called HCV, but are distinct enough to be referred to as HCV genotypes 1 (a or b), 2, 3, 4, 5, or 6 (e or o).
  participants
    Genotype 1a | 40 | 85 | 116 | 241
    Genotype 1b | 12 | 24 | 39 | 75
    Genotype 4 | 0 | 11 | 0 | 11
    Genotype 6 | 0 | 2 | 0 | 2
    Genotype 6e | 0 | 2 | 0 | 2
    Genotype 6o | 0 | 1 | 0 | 1
HCV RNA [Mean (Standard Deviation); unit: log10 copies/mL] | 6.5 (0.66) | 6.3 (0.73) | 6.4 (0.79) | 6.4 (0.75)
HCV RNA Category [Number; unit: participants]
  < 800,000 IU/mL | 7 | 33 | 28 | 68
  > 800,000 IU/mL | 45 | 92 | 127 | 264
Liver Biopsy Fibrosis Score [Number; unit: participants]
  Missing | 0 | 1 | 13 | 14
  Bridging Fibrosis | 7 | 17 | 23 | 47
  None or Minimal Fibrosis | 9 | 14 | 20 | 43
  Portal Fibrosis | 36 | 93 | 99 | 228
Alanine Aminotransferase (ALT) [Mean (Standard Deviation); unit: U/L] | 80.5 (71.61) | 83.7 (77.18) | 76.4 (55.91) | 79.8 (66.98)
ALT Category [Number; unit: participants] — The ULN for ALT was 60 IU/mL before March 26, 2012, then 56 IU/mL (males) and 45 IU/mL (females).
  participants
    ≤ 1.5 × the upper limit of the normal range (ULN) | 37 | 87 | 115 | 239
    > 1.5 × ULN | 15 | 38 | 40 | 93
IL28b Genotype [Number; unit: participants] — CC, CT, and TT alleles are different forms of the IL28b gene.
  participants
    CC | 13 | 36 | 39 | 88
    CT | 33 | 63 | 88 | 184
    TT | 6 | 26 | 28 | 60

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 24 Weeks Following Completion of Treatment (SVR24)
Description: SVR24 was defined as HCV RNA < the limit of detection (LOD; < 15 IU/mL) 24 weeks after the last dose of study drug.
Time Frame: Post-treatment Week 24
Population: Participants in the Safety Analysis Set (participants who were randomized and received at least 1 dose of study drug) with genotype 1 and who had available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF+PEG+RBV 12 Weeks | SOF+PEG+RBV 24 Weeks | SOF+PEG+RBV 12 Week/Rerandomization Group | SOF Rerandomization Group | SOF+RBV Rerandomization Group
Number analyzed (Participants) | 52 | 109 | 155 | 75 | 75
percentage of participants | 90.4 [79.0 to 96.8] | 92.7 [86.0 to 96.8] | 91.0 [85.3 to 95.0] | 93.3 [85.1 to 97.8] | 94.7 [86.9 to 98.5]
Statistical Analysis 1: Comparison: SOF+PEG+RBV 12 Weeks vs SOF+PEG+RBV 24 Weeks; The analyses was stratified by IL28B (CC versus any T allele) and plasma HCV RNA (< 800,000 IU/mL versus ≥ 800,000 IU/mL). Only participants with genotype 1 were included in the comparison due to the fact that participants with genotype 4 and 6 were only enrolled in the SOF+PEG+RBV 24 weeks group; Test type: Superiority or Other; p = 0.77, Cochran-Mantel-Haenszel — The p-value is based on the Cochran-Mantel-Haenszel (CMH) test stratified by randomization stratification factors; Difference in proportions = -1.4, 95% CI 2-sided [-12.2 to 9.4] — The difference in proportions and its 95% confidence interval (CI) were calculated based on stratum-adjusted Mantel-Haenszel (MH) proportions
Statistical Analysis 2: Comparison: SOF+PEG+RBV 12 Weeks vs SOF+PEG+RBV 12 Week/Rerandomization Group; The analyses was stratified by IL28B (CC versus any T allele) and plasma HCV RNA (< 800,000 IU/mL versus ≥ 800,000 IU/mL); Test type: Superiority or Other; p = 0.93, Cochran-Mantel-Haenszel — The p-value is based on the CMH test stratified by randomization stratification factors; The difference in proportions and its 95% CI were calculated based on stratum-adjusted MH proportions; Difference in proportions = -0.4, 95% CI 2-sided [-10.8 to 9.9]

2. Primary Outcome: Percentage of Participants Who Experienced Adverse Events
Description: Adverse events (AEs) occurring from baseline (Day 1 for all groups) to 30 days following the last dose of study drug were summarized across the participant population. A participant was counted once if they had a qualifying event.
Time Frame: Baseline (Day 1) to post-treatment Day 30
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF+PEG+RBV 12 Weeks | SOF+PEG+RBV 24 Weeks | SOF+PEG+RBV 12 Week/Rerandomization Group | SOF Rerandomization Group | SOF+RBV Rerandomization Group
Number analyzed (Participants) | 52 | 125 | 155 | 75 | 75
percentage of participants
  Any AE | 98.1 | 96.8 | 98.7 | 98.7 | 100.0
  Drug-related AE | 96.2 | 94.4 | 97.4 | 98.7 | 97.3
  Grade 3 or higher AE | 15.4 | 17.6 | 14.2 | 14.7 | 13.3
  AE leading to drug discontinuation | 5.8 | 16.0 | 4.5 | 5.3 | 4.0
  Serious AE | 3.8 | 4.8 | 2.6 | 2.7 | 2.7

3. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks Following Completion of Treatment (SVR12)
Description: SVR12 was defined as HCV RNA < LOD 12 weeks after the last dose of study drug.
Time Frame: Post-treatment Week 12
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF+PEG+RBV 12 Weeks | SOF+PEG+RBV 24 Weeks | SOF+PEG+RBV 12 Week/Rerandomization Group | SOF Rerandomization Group | SOF+RBV Rerandomization Group
Number analyzed (Participants) | 52 | 125 | 155 | 75 | 75
percentage of participants | 90.4 [79.0 to 96.8] | 92.0 [85.8 to 96.1] | 91.0 [85.3 to 95.0] | 93.3 [85.1 to 97.8] | 94.7 [86.9 to 98.5]

4. Secondary Outcome: Change in HCV RNA at Week 2
Time Frame: Baseline (Day 1) to Week 2
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF+PEG+RBV 12 Weeks | SOF+PEG+RBV 24 Weeks | SOF+PEG+RBV 12 Week/Rerandomization Group
Number analyzed (Participants) | 49 | 124 | 153
log10 IU/mL | -5.12 (0.660) | -5.07 (0.701) | -5.13 (0.768)

5. Secondary Outcome: Change in HCV RNA at Week 4
Time Frame: Baseline (Day 1) to Week 4
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF+PEG+RBV 12 Weeks | SOF+PEG+RBV 24 Weeks | SOF+PEG+RBV 12 Week/Rerandomization Group
Number analyzed (Participants) | 50 | 123 | 152
log10 IU/mL | -5.33 (0.649) | -5.19 (0.733) | -5.24 (0.785)

6. Secondary Outcome: Change in HCV RNA at Week 8
Time Frame: Baseline (Day 1) to Week 8
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF+PEG+RBV 12 Weeks | SOF+PEG+RBV 24 Weeks | SOF+PEG+RBV 12 Week/Rerandomization Group
Number analyzed (Participants) | 48 | 118 | 151
log10 IU/mL | -5.34 (0.635) | -5.17 (0.740) | -5.25 (0.789)

7. Secondary Outcome: Change in HCV RNA at Week 12
Time Frame: Baseline (Day 1) to Week 12
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF+PEG+RBV 12 Weeks | SOF+PEG+RBV 24 Weeks | SOF+PEG+RBV 12 Week/Rerandomization Group
Number analyzed (Participants) | 47 | 113 | 150
log10 IU/mL | -5.36 (0.616) | -5.20 (0.719) | -5.25 (0.791)

8. Secondary Outcome: Percentage of Participants With HCV RNA < LOD at Week 2
Time Frame: Week 2
Population: Participants in the Safety Analysis Set with Available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | SOF+PEG+RBV 12 Weeks | SOF+PEG+RBV 24 Weeks | SOF+PEG+RBV 12 Week/Rerandomization Group
Number analyzed (Participants) | 51 | 124 | 153
percentage of participants | 68.6 | 85.5 | 77.1

9. Secondary Outcome: Percentage of Participants With HCV RNA Below < LOD at Week 4
Time Frame: Week 4
Population: Participants in the Safety Analysis Set with Available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | SOF+PEG+RBV 12 Weeks | SOF+PEG+RBV 24 Weeks | SOF+PEG+RBV 12 Week/Rerandomization Group
Number analyzed (Participants) | 50 | 123 | 153
percentage of participants | 98.0 | 100.0 | 98.7

10. Secondary Outcome: Percentage of Participants With HCV RNA Below < LOD at Week 8
Time Frame: Week 8
Population: Participants in the Safety Analysis Set with Available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | SOF+PEG+RBV 12 Weeks | SOF+PEG+RBV 24 Weeks | SOF+PEG+RBV 12 Week/Rerandomization Group
Number analyzed (Participants) | 48 | 118 | 152
percentage of participants | 100.0 | 100.0 | 99.3

11. Secondary Outcome: Percentage of Participants With HCV RNA Below < LOD at Week 12
Time Frame: Week 12
Population: Participants in the Safety Analysis Set with Available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | SOF+PEG+RBV 12 Weeks | SOF+PEG+RBV 24 Weeks | SOF+PEG+RBV 12 Week/Rerandomization Group
Number analyzed (Participants) | 47 | 113 | 150
percentage of participants | 100.0 | 100.0 | 100.0

12. Secondary Outcome: Percentage of Participants With HCV RNA Below < LOD at Week 24
Time Frame: Week 24
Population: Participants in the Safety Analysis Set with Available data were analyzed. No participants in the SOF+PEG+RBV 12 weeks group were analyzed because they received only 12 weeks of treatment.
Measure: Number; unit: percentage of participants
Arm/Group | SOF+PEG+RBV 12 Weeks | SOF+PEG+RBV 24 Weeks | SOF Rerandomization Group | SOF+RBV Rerandomization Group
Number analyzed (Participants) | 0 | 100 | 68 | 74
percentage of participants |  | 100.0 | 100.0 | 98.6

13. Secondary Outcome: Percentage of Participants With ALT Normalization at Week 12
Description: ALT normalization was defined as ALT > ULN at baseline and ALT ≤ ULN at Week 12.
Time Frame: Baseline (Day 1) to Week 12
Population: Participants in the Safety Analysis Set with ALT > ULN at baseline and with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | SOF+PEG+RBV 12 Weeks | SOF+PEG+RBV 24 Weeks | SOF+PEG+RBV 12 Week/Rerandomization Group
Number analyzed (Participants) | 23 | 47 | 71
percentage of participants | 78.3 | 76.6 | 67.6

14. Secondary Outcome: Percentage of Participants With ALT Normalization at Week 24
Description: ALT normalization was defined as ALT > ULN at baseline (Day 1 for all groups) and ALT ≤ ULN at Week 24.
Time Frame: Baseline (Day 1) to Week 24
Population: Participants in the Safety Analysis Set with ALT > ULN at baseline and with available data were analyzed. No participants in the SOF+PEG+RBV 12 weeks group were analyzed because they received only 12 weeks of treatment.
Measure: Number; unit: percentage of participants
Arm/Group | SOF+PEG+RBV 12 Weeks | SOF+PEG+RBV 24 Weeks | SOF Rerandomization Group | SOF+RBV Rerandomization Group
Number analyzed (Participants) | 0 | 38 | 35 | 30
percentage of participants |  | 78.9 | 94.3 | 100.0

15. Secondary Outcome: Percentage of Participants With ALT Normalization at Post-treatment Week 4
Description: ALT normalization was defined as ALT > ULN at baseline (Day 1 for all groups) and ALT ≤ ULN at Post-treatment Week 4.
Time Frame: Baseline (Day 1) to Post-treatment Week 4
Population: Participants in the Safety Analysis Set with ALT > ULN at baseline and with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | SOF+PEG+RBV 12 Weeks | SOF+PEG+RBV 24 Weeks | SOF+PEG+RBV 12 Week/Rerandomization Group | SOF Rerandomization Group | SOF+RBV Rerandomization Group
Number analyzed (Participants) | 19 | 47 | 63 | 36 | 26
percentage of participants | 89.5 | 87.2 | 95.2 | 91.7 | 100.0

16. Secondary Outcome: Percentage of Participants With Virologic Failure During Treatment
Description: Virologic failure was defined as either
  * HCV RNA ≥ 15 IU/mL after having previously had HCV RNA < 15 IU/mL while on treatment, confirmed with 2 consecutive values or last available measurement (ie, breakthrough);
  * > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment, confirmed with 2 consecutive values or last available measurement (ie, rebound);or
  * HCV RNA persistently ≥ 15 IU/mL through 8 weeks of treatment (ie, nonresponse)
  Baseline was Day 1 for all groups.
Time Frame: Baseline (Day 1) to Week 24
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF+PEG+RBV 12 Weeks | SOF+PEG+RBV 24 Weeks | SOF+PEG+RBV 12 Week/Rerandomization Group | SOF Rerandomization Group | SOF+RBV Rerandomization Group
Number analyzed (Participants) | 52 | 125 | 155 | 75 | 75
percentage of participants
  Viral breakthrough | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Viral rebound | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Non-response | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

17. Secondary Outcome: Percentage of Participants With Virologic Failure Following Treatment (Viral Relapse).
Description: Viral relapse was defined as HCV RNA < 15 IU/mL at end of treatment, confirmed with 2 consecutive values or last available measurement.
Time Frame: End of treatment to Post-treatment Week 24
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | SOF+PEG+RBV 12 Weeks | SOF+PEG+RBV 24 Weeks | SOF+PEG+RBV 12 Week/Rerandomization Group | SOF Rerandomization Group | SOF+RBV Rerandomization Group
Number analyzed (Participants) | 51 | 124 | 153 | 75 | 75
percentage of participants | 5.9 | 1.6 | 3.9 | 2.7 | 2.7

ADVERSE EVENTS:
Time Frame: Baseline (Day 1) to Week 12 or Week 24 (depending upon treatment arm) plus 30 days. Adverse events are counted if they began on or after the date of the first dose and on or before the last dose of study drug plus 30 days.
Description: As prespecified in the analysis plan, adverse events are reported according to the group to which participants were initially randomized.
Arm/Group | SOF+PEG+RBV 12 Weeks | SOF+PEG+RBV 24 Weeks | SOF+PEG+RBV 12 Week/Rerandomization Group
Serious Adverse Events (participants affected / at risk) | 2/52 | 6/125 | 4/155
Other Adverse Events (participants affected / at risk) | 51/52 | 121/125 | 153/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOF+PEG+RBV 12 Weeks (N=52) | SOF+PEG+RBV 24 Weeks (N=125) | SOF+PEG+RBV 12 Week/Rerandomization Group (N=155)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 0
Colitis iscaemic (Gastrointestinal disorders) | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 0 | 1
Chelocystitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1 | 0
Alcoohol poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Hip arthroplasty (Surgical and medical procedures) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SOF+PEG+RBV 12 Weeks (N=52) | SOF+PEG+RBV 24 Weeks (N=125) | SOF+PEG+RBV 12 Week/Rerandomization Group (N=155)
Anaemia (Blood and lymphatic system disorders) | 7 | 31 | 34
Neutropenia (Blood and lymphatic system disorders) | 12 | 25 | 22
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 0 | 3
Vision blurred (Eye disorders) | 6 | 6 | 6
Nausea (Gastrointestinal disorders) | 16 | 43 | 51
Diarrhoea (Gastrointestinal disorders) | 11 | 23 | 20
Vomiting (Gastrointestinal disorders) | 3 | 17 | 18
Constipation (Gastrointestinal disorders) | 3 | 6 | 12
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 8 | 8
Dry mouth (Gastrointestinal disorders) | 1 | 8 | 7
Abdominal pain upper (Gastrointestinal disorders) | 3 | 3 | 7
Abdominal pain (Gastrointestinal disorders) | 1 | 7 | 4
Flatulence (Gastrointestinal disorders) | 4 | 2 | 0
Fatigue (General disorders) | 25 | 63 | 86
Chills (General disorders) | 15 | 25 | 29
Pyrexia (General disorders) | 18 | 15 | 26
Pain (General disorders) | 9 | 14 | 24
Irritability (General disorders) | 6 | 15 | 14
Influenza like illness (General disorders) | 3 | 10 | 14
Injection site erythemia (General disorders) | 4 | 6 | 10
Injection site reaction (General disorders) | 3 | 5 | 9
Asthenia (General disorders) | 3 | 7 | 4
Injection site rash (General disorders) | 0 | 4 | 8
Upper respiratory tract infection (Infections and infestations) | 1 | 7 | 8
Urinary tract infection (Infections and infestations) | 0 | 6 | 10
Nasopharyngitis (Infections and infestations) | 2 | 3 | 9
Sinusitis (Infections and infestations) | 1 | 7 | 4
Decreased appetite (Metabolism and nutrition disorders) | 7 | 17 | 34
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 | 23 | 14
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 17 | 23
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 11 | 12
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 12 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 6 | 8
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 6 | 5
Headache (Nervous system disorders) | 14 | 38 | 65
Dizziness (Nervous system disorders) | 8 | 19 | 21
Dysgeusia (Nervous system disorders) | 3 | 3 | 10
Disturbance in attention (Nervous system disorders) | 1 | 4 | 9
Insomnia (Psychiatric disorders) | 12 | 28 | 36
Anxiety (Psychiatric disorders) | 4 | 17 | 22
Depression (Psychiatric disorders) | 4 | 17 | 19
Affect lability (Psychiatric disorders) | 4 | 4 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 18 | 21
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 11 | 22
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 6
Rash (Skin and subcutaneous tissue disorders) | 7 | 26 | 39
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 18 | 16
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 15 | 10
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 9 | 7
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 8 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years